CLINICAL TRIAL: NCT06873802
Title: ZTE MRI Pulse Sequence Use for Visualization of Bone Cement, Breast Biopsy Markers
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Sponsor
Other Study IDs: 24-010877; NCI-2025-01494 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 24-010877 (Other: Mayo Clinic Institutional Review Board); R01EB033008 (NIH)
Record Dates: First submitted 2025-03-11; First posted 2025-03-13 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational: Participants undergo standard of care MRI breast imaging with conventional or bone cement breast biopsy markers and complete a questionnaire on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study is being done to determine if a clinically available MRI sequence called ZTE imaging better visualizes breast biopsy markers made of bone cement compared to the currently used breast biopsy markers made of metal.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To demonstrate that clinically available ZTE imaging allows for better visualization of bone cement breast biopsy markers when compared to conventional breast biopsy markers and pulse sequences.

OUTLINE: This is an observational study.

Participants undergo standard of care MRI breast imaging with conventional or bone cement breast biopsy markers and complete a questionnaire on study.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 or older

Exclusion Criteria:

* Cardiac pacemaker
* Implanted cardiac defibrillator
* Internal pacing wires
* Cerebral, carotid, or aortic aneurysmal clips
* Cochlear implants
* Implanted tissue expanders
* Claustrophobia
* Cannot lay prone

  * Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy individuals that can receive a non-contrast enhanced breast MRI
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2025-04-11 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-25 (Actual)

PRIMARY OUTCOMES:
Bone cement marker (BCM) images compared to conventional images | Baseline
  Will be assessed using zero echo-time (ZTE) and standard breast biopsy pulse sequences. Two radiologists will interpret images, evaluating the pulse sequences and ZTE images for marker conspicuity. Each sequence will receive a score for conspicuity ranging from 0 to 2. A score of 0 indicates 'not seen, 1 'maybe seen,' and 2 'well seen.'

CONTACTS AND LOCATIONS:
Overall Officials: Christine U. Lee, MD, PhD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

DOCUMENTS (1):
  • Informed Consent Form (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/02/NCT06873802/ICF_000.pdf